CLINICAL TRIAL: NCT04964258
Title: A Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-105 in Healthy Subjects
Brief Title: A Study of TAK-105 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: TAK-105-1001
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1: Placebo (Placebo Comparator): TAK-105-a matching-placebo, injection, subcutaneously, once on Day 1.
  Interventions: Drug: TAK-105-a Placebo
- Part 1: TAK-105 Dose 1 (Experimental): TAK-105-a Dose 1, injection, subcutaneously, once on Day 1.
  Interventions: Drug: TAK-105-a
- Part 1: TAK-105 Dose 2 (Experimental): TAK-105-a Dose 2, injection, subcutaneously, once on Day 1.
  Interventions: Drug: TAK-105-a
- Part 1: TAK-105 Dose 3 (Experimental): TAK-105-a Dose 3, injection, subcutaneously, once on Day 1.
  Interventions: Drug: TAK-105-a
- Part 1: TAK-105 Dose 4 (Experimental): TAK-105-a Dose 4, injection, subcutaneously, once on Day 1.
  Interventions: Drug: TAK-105-a
- Part 1: TAK-105 Dose 5 (Experimental): TAK-105-a Dose 5, injection, subcutaneously, once on Day 1.
  Interventions: Drug: TAK-105-a
- Part 1: TAK-105 Dose 6 (Experimental): TAK-105-a Dose 6, injection, subcutaneously, once on Day 1.
  Interventions: Drug: TAK-105-a
- Part 1: TAK-105 Dose 7 (Experimental): TAK-105-a Dose 7, injection, subcutaneously, once on Day 1.
  Interventions: Drug: TAK-105-a
- Part 2: Placebo (Placebo Comparator): TAK-105-a matching-placebo, injection, subcutaneously, once weekly for 4 weeks.
  Interventions: Drug: TAK-105-a Placebo
- Part 2: TAK-105 Dose 1A (Experimental): TAK-105-a Dose 1A, injection, subcutaneously, once weekly for up to 4 weeks.
  Interventions: Drug: TAK-105-a
- Part 2: TAK-105 Dose 2A (Experimental): TAK-105-a Dose 2A, injection, subcutaneously, once weekly for 1 week.
  Interventions: Drug: TAK-105-a

INTERVENTIONS:
Drug: TAK-105-a — TAK-105-a subcutaneous solution.
  Arms: Part 1: TAK-105 Dose 1; Part 1: TAK-105 Dose 2; Part 1: TAK-105 Dose 3; Part 1: TAK-105 Dose 4; Part 1: TAK-105 Dose 5; Part 1: TAK-105 Dose 6; Part 1: TAK-105 Dose 7; Part 2: TAK-105 Dose 1A; Part 2: TAK-105 Dose 2A
Drug: TAK-105-a Placebo — TAK-105-a placebo-matching solution.
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
It is hoped that in the future, TAK-105 will be used to help treat people with nausea and vomiting. The main aims of this study are as follows:

* To check for side effects from TAK-105 in healthy adults.
* To learn how much TAK-105 they can receive without getting side effects from it.

Participants will receive either TAK-105 as TAK-105-a or TAK-105-b (depending upon the part they are enrolled in) or a placebo as an injection under the skin (sub-cutaneous injection). A placebo looks like TAK-105-a or TAK-105-b but will not have any medicine in it. Three times as many participants will receive TAK-105-a or TAK-105-b than placebo.

The study will have 6 parts. Each part will have several small groups of participants, called cohorts. Participants will only be in 1 cohort in 1 part of the study.

Part 1: Participants will check into the study clinic to receive a single dose of TAK-105-a or placebo and will stay in the clinic for about 10 days. Then, participants return to the clinic for follow-up visits up to about 60 days after the dose.

Part 2: Participants will check into the study clinic to receive TAK-105-a or placebo once a week for 4 weeks, and will stay in the clinic for about 26 days. Then, participants return to the clinic for follow-up visits up to about 60 days after last dose.

Part 3: Participants will check into the study clinic to receive 2, 3 or 4 weekly doses of TAK-105-a or placebo. Their clinic stay will be for 10 to 24 days depending which cohort they are in. Then, participants return to the clinic for follow-up visits up to about 28 days after last dose.

Part 4: Participants will check into the study clinic to receive 2 doses (once a week for 2 weeks) of TAK-105-a or placebo and will stay in the study clinic for about 12 days. They will return to the clinic later (in about 1-3 weeks) for another (third) dose and will stay for 2 days after the third dose. Then, participants return to the clinic for follow-up visits up to about 3 months after first dose.

Part 5a: Participants will check into the study clinic to receive a single dose of TAK-105-a or placebo and will stay in the clinic for about 10 days. Then, participants return to the clinic for follow-up visits up to about 60 days after the dose.

Part 5b: Participants will check into the study clinic to receive TAK-105-a or placebo once a week for 4 weeks, and will stay in the clinic for about 26 days. Then, participants return to the clinic for follow-up visits up to about 60 days after last dose. Part 5b will be optional, depending on the pharmacokinetic (PK) and safety data observed in Part 2.

Part 6: Participants will check into the study clinic to receive a single dose of TAK-105-b or placebo and will stay in the clinic for about 10 days. Then, participants return to the clinic for follow-up visits up to about 60 days after the dose.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-105. The study will look at the safety, tolerability, and PK of TAK-105-a and TAK-105-b in healthy participants.

Participants in each cohort will be randomized to receive treatment with TAK-105-a or TAK-105-b or matching placebo which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need). The study consists of 6 parts and up to 34 cohorts as mentioned below:

* Part 1 (SRD) will enroll healthy participants in up to 12 cohorts.
* Part 2 (MRD) will enroll healthy participants in up to 5 ascending cohorts.
* Part 3 (Dose titration) will enroll healthy participants in up to 6 multiple-dose cohorts.
* Part 4 (Redosing) will enroll healthy participants in up to 4 redosing cohorts.
* Part 5a (SRD) will enroll healthy Japanese participants in up to 3 cohorts.
* Part 5b (MRD) (optional) will enroll healthy Japanese participants in up to 2 cohorts. The MRD cohorts in Part 5b will be optional, depending on the PK and safety data observed in Part 2 (MRD).
* Part 6 (SRD) will enroll healthy participants in up to 2 cohorts.

Each cohort in all the parts will have 8 randomized participants with 6 participants receiving a single dose of TAK-105-a in Parts 1 to 5 or TAK-105-b in Part 6, and 2 receiving TAK-105-a matching placebo (Parts 1 to 5) or TAK-105-b matching placebo (Part 6) in a 3:1 ratio. This multi-center trial will be conducted in the United States. The overall duration of the study is approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

For All Cohorts

1. Must have a body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 30.0 kilogram per square meter (kg/m^2).
2. Continuous nonsmoker who has not used nicotine and tobacco-containing products for at least 3 months prior to screening and through discharge.
3. Be judged to be in good health (example, no evidence of psychiatric, hepatic, renal, pulmonary, or cardiovascular disease) by the investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, electrocardiogram (ECG), and vital sign measurements performed at the screening visit and before administration of the initial dose of study drug or invasive procedure.

   For Japanese participants in Part 5 (Cohorts 28 to 32 only):
4. Has 2 Japanese parents and 4 Japanese grandparents, as confirmed by interview.

Exclusion Criteria:

1. Participated in another investigational study within 4 weeks (or based on local regulations) or within 5 half-lives of the investigational product before the screening visit. The 4-week or 5 half-lives window will be derived from the date of the last dose and/or adverse event (AE) related to the study procedure in the previous study to the screening visit of the current study.
2. Has a history of significant multiple and/or severe allergies (example, food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance to prescription or nonprescription drugs or food.
3. Has a known hypersensitivity or contraindication to any component of TAK 105.
4. Has positive pregnancy test or is lactating or breastfeeding.
5. Has known or suspected current coronavirus disease 2019 (COVID-19) infection or is at risk of COVID-19 infection as assessed by the investigator.
6. Unable to refrain from or anticipates using all medications including herbal medicines beginning approximately 7 days before administration of the first dose of study drug, throughout the study until the last follow-up visit.
7. With history or presence of:

   * 3 or more incidences of syncope (example, vasovagal) within the last 5 years prior to screening;
   * A family history of unexplained sudden death or channelopathy;
   * Brugada syndrome (RBBB [right bundle branch block] pattern with ST-elevation in leads V1 V3);
   * CV or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction, stroke, sick sinus syndrome, pulmonary congestion, symptomatic or significant cardiac arrhythmia, supraventricular or ventricular tachycardia, second-degree atrioventricular (AV) block type 2, third degree AV block, prolonged QT interval with Fridericia correction method (QTcF) interval, hypokalemia, hypomagnesemia, or conduction abnormalities;
   * Risk factors for Torsade de Pointes (example, heart failure, cardiomyopathy, or family history of Long QT Syndrome);
   * Any clinically significant ECG findings or medical history including: long or short QTcF (over 450 milli second [msec] or less than 360 msec), bifascicular block or QRS greater than equal to (>=)120 msec or PR interval > 200 msec at screening or Day 1 pre-Hour 0;
   * Has a documented history of sinus bradycardia less than (<) 45 beats per minute [bpm]) based upon vital signs assessments, sinoatrial block as evidenced on ECG or sinus pause >=3 seconds on ECG or predose telemetry.
8. Has an average semi recumbent blood pressure (BP) less than 90 (systolic) and 60 (diastolic) millimeter of mercury (mmHg) or greater than 140/90 mmHg from screening to predose, inclusive.
9. From screening to Day -2, participants with an average semirecumbent heart rate (HR) <55 or >100 beats per minute (bpm) should be excluded. From Day -2 to predose, enrollment of participants with an average HR <55 or >100 bpm will be left to the judgment of the investigator, unless HR is <50 bpm, which must be discussed with the medical monitor for approval.
10. Has orthostatic hypotension defined as a decrease in systolic BP (SBP) >=20 mmHg or a decrease in diastolic BP (DPB) >=10 mmHg at approximately 2 minutes of standing when compared with BP from the semirecumbent position at screening to predose assessments, inclusive.
11. Has postural orthostatic tachycardia, defined as an increase of >30 bpm or HR >120 bpm at approximately 2 minutes of standing, at screening to predose assessments, inclusive.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- United States (3):
  - Celerion, Tempe, Arizona
  - PPD Development, LP, Las Vegas, Nevada
  - PPD Development, LP, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click on this link. — https://clinicaltrials.takeda.com/study-detail/60f5c5d0f883ca001e82d354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants took part in the study at 3 investigative sites in the United States from 26 July 2021 to 20 June 2023. The study consisted of six parts: Participants were enrolled into Part 1 and Part 2 of the study. Study was completed after Parts 1 and 2. Sponsor decided not to conduct Part 3, 4, 5, and 6 after comprehensive review of available data.
Pre-assignment Details: Participants were randomized in Parts 1 and 2 to receive of either TAK-105 or matching-placebo.
Groups:
- Part 2: TAK-105 Dose 1A: TAK-105-a Dose 1A, injection, subcutaneously, once weekly for 2 and 4 weeks.
Period: Overall Study
Arm/Group | Part 1: Placebo | Part 1: TAK-105 Dose 1 | Part 1: TAK-105 Dose 2 | Part 1: TAK-105 Dose 3 | Part 1: TAK-105 Dose 4 | Part 1: TAK-105 Dose 5 | Part 1: TAK-105 Dose 6 | Part 1: TAK-105 Dose 7 | Part 2: Placebo | Part 2: TAK-105 Dose 1A | Part 2: TAK-105 Dose 2A
Started | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6
Completed | 13 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 12 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were randomized and received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: TAK-105 Dose 1 | Part 1: TAK-105 Dose 2 | Part 1: TAK-105 Dose 3 | Part 1: TAK-105 Dose 4 | Part 1: TAK-105 Dose 5 | Part 1: TAK-105 Dose 6 | Part 1: TAK-105 Dose 7 | Part 2: Placebo | Part 2: TAK-105 Dose 1A | Part 2: TAK-105 Dose 2A | Total
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 3 | 0 | 12
  Male | 13 | 5 | 5 | 6 | 5 | 5 | 6 | 4 | 4 | 9 | 6 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 3 | 3 | 3 | 3 | 1 | 2 | 4 | 8 | 5 | 42
  Not Hispanic or Latino | 7 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 2 | 4 | 1 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 1 | 1 | 1 | 4 | 3 | 2 | 0 | 1 | 0 | 18
  White | 10 | 5 | 5 | 5 | 4 | 2 | 3 | 4 | 5 | 11 | 5 | 59
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With At Least One Treatment-emergent Adverse Event (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an AE that started or worsened after the first dose of the study treatment and last dose of study treatment.
Time Frame: Part 1: Baseline up to Day 60; Part 2: Baseline up to Day 82
Population: Safety analysis set included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: TAK-105 Dose 1 | Part 1: TAK-105 Dose 2 | Part 1: TAK-105 Dose 3 | Part 1: TAK-105 Dose 4 | Part 1: TAK-105 Dose 5 | Part 1: TAK-105 Dose 6 | Part 1: TAK-105 Dose 7 | Part 2: Placebo | Part 2: TAK-105 Dose 1A | Part 2: TAK-105 Dose 2A
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6
Participants | 6 | 3 | 4 | 3 | 4 | 3 | 5 | 4 | 6 | 9 | 6

2. Secondary Outcome: Number of Participants Based on Antidrug Antibody (ADA) Status
Description: ADA included ADA-negative or transiently and persistently ADA-positive, and low or high ADA titer assessment. ADA negative was defined as participants who did not have a confirmed positive ADA status in any postbaseline assessment. Transiently ADA positive was defined as participants who had confirmed positive ADA status in 1 or 2 postbaseline assessments. Persistently ADA positive was defined as participants who had confirmed positive ADA status in more than 2 postbaseline assessments. For ADA positive (transiently ADA positive or persistently ADA positive) only, high ADA titer was defined as participant who has at least 1 postbaseline ADA titer greater than (>) 16; low ADA titer was defined as participant whose postbaseline ADA titers were all less than or equal to (<=) 16. ADA titer was assessed in ADA-positive participants.
Time Frame: Part 1: Baseline up to Day 60; Part 2: Baseline up to Day 82
Population: Immunogenicity analysis set included all participants who received at least 1 dose of study treatment and had the baseline sample and at least 1 postbaseline sample ADA assessment. Here, "number analyzed" signifies participants who were evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: TAK-105 Dose 1 | Part 1: TAK-105 Dose 2 | Part 1: TAK-105 Dose 3 | Part 1: TAK-105 Dose 4 | Part 1: TAK-105 Dose 5 | Part 1: TAK-105 Dose 6 | Part 1: TAK-105 Dose 7 | Part 2: Placebo | Part 2: TAK-105 Dose 1A | Part 2: TAK-105 Dose 2A
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6
Participants
  ADA Negative | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6
  Persistently ADA Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Transiently ADA Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA Titer Low: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA Titer High: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Parts 1, and 2, Cmax: Maximum Observed Plasma Concentration for TAK-105
Description: Due to confidentiality reasons and chances of exposing the doses for TAK-105, the data for this pharmacokinetic outcome measure was not reported.
Time Frame: Part 1: Day 1 pre-dose and at multiple timepoints (up to Day 60) post-dose; Part 2: Day 1 pre-dose and at multiple timepoints (up to Day 6) post-dose; Part 2: Day 22 pre-dose and at multiple timepoints (up to Day 82) post-dose
Population: PK analysis set included all participants who received at least 1 dose of TAK-105 and had at least 1 measurable post-dose plasma or urine concentration for TAK-105. As per-planned analysis, for PK assessment, participants in the Dose 1A arm group were divided and analyzed into two separate groups based on the number of Dose 1A doses received (i.e., who received all 4 doses' and 'who received 2 doses).
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Part 1, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-105
Description: as for outcome 3
Time Frame: Part 1: Day 1 pre-dose and at multiple timepoints (up to Day 60) post-dose
Population: PK analysis set. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Data was not planned to be analyzed for Part 2
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Parts 1, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-105
Description: as for outcome 3
Time Frame: Part 1: Day 1 pre-dose and at multiple timepoints (up to Day 60) post-dose
Population: PK analysis set. Data was not planned to be analyzed for Part 2.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Parts 1, and 2, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-105
Description: as for outcome 3
Time Frame: as for outcome 3
Population: PK analysis set. As per-planned analysis, for PK assessment, participants in the Dose 1A arm group were divided and analyzed into two separate groups based on the number of Dose 1A doses received (i.e., who received all 4 doses' and 'who received 2 doses).
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Parts 1, and 2, T1/2z: Terminal Disposition Phase Half-life for TAK-105
Description: as for outcome 3
Time Frame: as for outcome 3
Population: PK analysis set. As per-planned analysis, for PK assessment, participants in the Dose 1A arm group were divided and analyzed into two separate groups based on the number of Dose 1A doses received (i.e., who received all 4 doses' and 'who received 2 doses). Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Parts 1, and 2, CL/F: Apparent Clearance After Extravascular Administration for TAK-105
Description: as for outcome 3
Time Frame: Part 1: Day 1 pre-dose and at multiple timepoints (up to Day 60) post-dose; Part 2: Day 22 pre-dose and at multiple timepoints (up to Day 82) post-dose
Population: as for outcome 7
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Parts 1, and 2, Vz/F: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration for TAK-105
Description: as for outcome 3
Time Frame: as for outcome 8
Population: as for outcome 7
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Part 2, AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to Tau Over Dosing Interval for TAK-105
Description: as for outcome 3
Time Frame: Part 2: Day 1 pre-dose and at multiple timepoints (up to Day 6) post-dose; Day 22 pre-dose and at multiple timepoints (up to Day 82) post-dose
Population: PK analysis set. Data was not planned to be analyzed for Part 1. As per-planned analysis, for PK assessment, participants in the Dose 1A arm group were divided and analyzed into two separate groups based on the number of Dose 1A doses received (i.e., who received all 4 doses' and 'who received 2 doses). Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Part 2, Ctrough: Observed Plasma Concentration at the End of a Dosing Interval at Steady State for TAK-105
Description: as for outcome 3
Time Frame: Part 2: Day 22 pre-dose and at multiple timepoints (up to Day 82) post-dose
Population: as for outcome 10
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Parts 1, and 2, Aet: Amount of Drug Excreted in Urine From Time 0 to Time t for TAK-105
Description: as for outcome 3
Time Frame: Parts 1 and 2: Day 1 pre-dose and at multiple time points (up to Day 8) post-dose; Part 2: Day 22 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: PK analysis set. As per-planned analysis, for PK assessment, participants in the Dose 1A arm group were divided and analyzed into two separate groups based on the number of Dose 1A doses received (i.e., Who received all 4 doses' and 'who received 2 doses). Here, "overall number of participants analyzed" signifies participants evaluable for this outcome. Data of urine PK parameter could not be calculated as all samples were below the lower limit of quantification (LLOQ) values in Parts 1 and 2.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Parts 1, and 2, Aet1-t2: Amount of Drug Excreted in Urine From Time 1 to Time 2 for TAK-105
Description: as for outcome 3
Time Frame: as for outcome 12
Population: PK analysis set. As per-planned analysis, for PK assessment, participants in the Dose 1A arm group were divided and analyzed into two separate groups based on the number of Dose 1A doses received (i.e., Who received all 4 doses' and 'who received 2 doses). Here, "overall number of participants analyzed" signifies participants evaluable for this outcome. Data of urine PK parameter could not be calculated as all samples were below the LLOQ values in Parts 1 and 2.
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Parts 1, and 2, Aeτ: Amount of Drug Excreted in Urine During a Dosing Interval (τ) at Steady State for TAK-105
Description: as for outcome 3
Time Frame: as for outcome 12
Population: as for outcome 13
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Parts 1, and 2, fe,t: Fraction of Administered Dose of Drug Excreted From Urine From Time 0 to Time t for TAK-105
Description: as for outcome 3
Time Frame: as for outcome 12
Population: as for outcome 13
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Parts 1, and 2, CLR: Renal Clearance for TAK-105
Description: as for outcome 3
Time Frame: as for outcome 12
Population: as for outcome 13
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Part 1: Baseline up to Day 60; Part 2: Baseline up to Day 82
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1: Placebo | Part 1: TAK-105 Dose 1 | Part 1: TAK-105 Dose 2 | Part 1: TAK-105 Dose 3 | Part 1: TAK-105 Dose 4 | Part 1: TAK-105 Dose 5 | Part 1: TAK-105 Dose 6 | Part 1: TAK-105 Dose 7 | Part 2: Placebo | Part 2: TAK-105 Dose 1A | Part 2: TAK-105 Dose 2A
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6 | 1/6 | 0/6 | 0/6 | 0/6 | 1/6 | 1/6 | 1/6 | 1/12 | 1/6
Other Adverse Events (participants affected / at risk) | 6/14 | 3/6 | 4/6 | 3/6 | 4/6 | 3/6 | 4/6 | 4/6 | 5/6 | 9/12 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=14) | Part 1: TAK-105 Dose 1 (N=6) | Part 1: TAK-105 Dose 2 (N=6) | Part 1: TAK-105 Dose 3 (N=6) | Part 1: TAK-105 Dose 4 (N=6) | Part 1: TAK-105 Dose 5 (N=6) | Part 1: TAK-105 Dose 6 (N=6) | Part 1: TAK-105 Dose 7 (N=6) | Part 2: Placebo (N=6) | Part 2: TAK-105 Dose 1A (N=12) | Part 2: TAK-105 Dose 2A (N=6)
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=14) | Part 1: TAK-105 Dose 1 (N=6) | Part 1: TAK-105 Dose 2 (N=6) | Part 1: TAK-105 Dose 3 (N=6) | Part 1: TAK-105 Dose 4 (N=6) | Part 1: TAK-105 Dose 5 (N=6) | Part 1: TAK-105 Dose 6 (N=6) | Part 1: TAK-105 Dose 7 (N=6) | Part 2: Placebo (N=6) | Part 2: TAK-105 Dose 1A (N=12) | Part 2: TAK-105 Dose 2A (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Medical device site dermatitis (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 6
Medical device site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Medical device site irritation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Medical device site papule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Medical device site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Medical device site vesicles (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 1 | 2 | 1 | 3 | 2 | 3 | 2 | 1 | 5 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT04964258/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT04964258/SAP_001.pdf